CLINICAL TRIAL: NCT03545776
Title: Teaching the Basics of Electroencephalography to Critical Care Teams
Brief Title: Critical Care EEG Course
Status: Completed | Type: Observational
Sponsor: Ictal Group (Other)
Collaborators: Versailles Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Critical Care EEG Course
Record Dates: First submitted 2018-05-07; First posted 2018-06-04 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Electroencephalogram; Intensive Care Units; Teaching Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Educational program: Medical and nursing staff will be given a 10-points EEG face-to-face initial training course that will be preceded by a pre-test evaluation and followed by delayed post-test evaluations.
  Training will be followed by an online teaching consisting on additional questions and answers quizzes based on the 10 educational goals already described elsewhere.
  In order to avoid any risk of intrasite contamination, all the learners benefiting from the training in the same department will be trained in a uniform time, with respect to the training schedule regarding post-test evaluations (day-1, day-15 and day-30). A final evaluation will be performed at day-90 after beginning of the training course.
  Interventions: Other: Critical Care EEG Course

INTERVENTIONS:
Other: Critical Care EEG Course — Medical and nursing staff will be given a 10-points EEG face-to-face initial training course followed by an online teaching and educational quizzes at day-1, day-15 and day-30 after initial training. A final evaluation will be performed at day-90 after beginning of the training course.
  10-points EEG educational objectives : physiological rhythms, reactivity, symmetry, effects of sedation, burst suppression, paroxysmal activities, periodic / pseudoperiodic activities, rhythmic activities, artifacts, null EEG

SUMMARY:
Knowledge of the basic fundamental skills of electroencephalography would enable medical and nursing staffs to provide efficient and effective bedside EEG monitoring in critically ill patients.

The aim of this study is to evaluate the ability of a 10-points EEG teaching program to allow bedside caregivers (medical and nursing intensive care unit staff) interpreting EEG in the critical care setting.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers among medical and nursing ICU staff of the participating ICUs

Exclusion Criteria:

* Experienced or trained ICU staff members to EEG interpretation (pre-test score > 5/10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critical care medical and nursing staff
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Overall EEG interpretation | at Day 90
  Percentage of learners with a correct answer rate.Training will be considered as efficient if more than 75% of learners are associated with a correct answer rate above 80% to EEG interpretation test at day 90 after initial training.

SECONDARY OUTCOMES:
Before/After Comparison | from Day 1 to Day 90 after face-to-face training
  Comparison of correct answer rate between pre-test and post-tests evaluations at day 1, day 15, day 30 and day 90 after face-to-face training Analyzes will be carried out according to each of the 10-points educational goals, according to the medical or nursing staff category, according to the student's degree and according to the center and to usual way of using EEG (continuous, sequential, external provider)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Medico-Surgical Intensive Care Unit - Ambroise Pare Hospital, Boulogne-Billancourt
  - Department of Anesthesia and Critical Care, Beaujon Hospital, Clichy
  - Intensive Care Unit - Versailles Hospital, Le Chesnay
  - Medical Intensive Care Unit - Cochin Teaching Hospital, Paris
  - Medico-Surgical Intensive Care Unit - Saint Joseph Hospital, Paris
  - Intensive Care Unit - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legriel S, Jacq G, Lalloz A, Geri G, Mahaux P, Bruel C, Brochon S, Zuber B, Andre C, Dervin K, Holleville M, Cariou A. Teaching Important Basic EEG Patterns of Bedside Electroencephalography to Critical Care Staffs: A Prospective Multicenter Study. Neurocrit Care. 2021 Feb;34(1):144-153. doi: 10.1007/s12028-020-01010-5. PMID 32495314